CLINICAL TRIAL: NCT05001737
Title: A Two-cohort, Open-label, Single Arm, Multicenter Study to Evaluate Efficacy, Safety and Tolerability, PK and PD, of Emapalumab in Children and Adults With MAS in Still's Disease or With MAS in Systemic Lupus Erythematous
Brief Title: Evaluate Efficacy, Safety and Tolerability, PK and PD of Emapalumab in Children and Adults With MAS in Still's or SLE
Acronym: EMERALD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Swedish Orphan Biovitrum (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NI-0501-14; 2021-001577-24 (EudraCT Number)
Record Dates: First submitted 2021-06-16; First posted 2021-08-12 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Macrophage Activation Syndrome; Secondary Hemophagocytic Lymphohistiocytosis; Still Disease; Systemic Lupus Erythematosus; SJIA; AOSD; MAS
MeSH Terms: conditions — Macrophage Activation Syndrome; Arthritis, Juvenile; Lupus Erythematosus, Systemic | interventions — Emapalumab; World Health Organization

STUDY DESIGN:
Intervention Model Description: 2 cohorts
Masking Description: Open label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Cohort 1 (sJIA and AOSD) and Cohort 2 (SLE) (Experimental): MAS in the context of systemic juvenile idiopathic arthritis and adult onset Still's disease (sJIA and AOSD) or SLE
  Interventions: Drug: Emapalumab

INTERVENTIONS:
Drug: Emapalumab — Emapalumab iv infusion
  Other Names: NI-0501; emapalumab-lzsg; ATC code: L04AA39 (WHO)

SUMMARY:
The purpose of this study is to assess the safety, tolerability and efficacy of emapalumab in children and adults with macrophage activation syndrome (sHLH/MAS) in Still's disease (including systemic juvenile idiopathic arthritis and adult onset Still's disease) or with sHLH/MAS in systemic lupus erythematous, resenting an inadequate response to high dose glucocorticoid treatment.

DETAILED DESCRIPTION:
Study NI-0501-14 is a two-cohort trial that enrolls subjects who are diagnosed with sHLH/MAS (MAS being a form of secondary HLH) and who are presenting an inadequate response to high doses of GCs. These subjects will be enrolled in 2 cohorts as per their background disease. The cohorts are defined as follows:

* Cohort 1: MAS in the context of sJIA and AOSD.
* Cohort 2: MAS in the context of pediatric and adult SLE.

The study has the objectives to investigate the efficacy, safety and tolerability, for 8 weeks, and PK and PD, QoL and immunogenicity in these 2 cohorts for up to 1 year after last dose of of emapalumab.

Macrophage Activation Syndrome (MAS) Secondary Hemophagocytic Lymphohistiocytosis (sHLH) systemic Juvenile Idiopathic Arthritis (sJIA) Adult-onset Still's Disease (AOSD) Systemic Lupus Erythematosus (SLE)

ELIGIBILITY:
Inclusion criteria Run-in phase in all cohorts

1. Informed consent provided by the subject or by the subject s' legally authorized representative(s) with the assent of subjects who are legally capable of providing it, as required by local law.
2. Male and female subjects aged between 6 months and 80 years of age at the time of diagnosis of MAS.
3. MAS defined as per the criteria defined below for each cohort and requiring treatment with GCs.

Interventional phase in all cohorts

1. Informed consent provided by the subject or by the subject's legally authorized representative(s) with the assent of subjects who are legally capable of providing it, as as required by local law.
2. Male and female subjects aged between 6 months and 80 years of age at the time of diagnosis of active MAS.
3. Subjects who have shown an inadequate response to high dose intravenous (i.v.) GCs administered for at least 3 days according to local standard clinical practice, including but not limited to pulses of 30 mg/kg PDN on 3 consecutive days. High i.v. GCs dose is recommended not to be lower than 2 mg/kg/ day PDN equivalent (or at least 60 mg/day in pediatric subjects of 30 kg or more, and at least 1g/day in adult MAS subjects). In case of rapid worsening of the subject's condition and/or laboratory parameters, as per Investigator judgment, inclusion may occur within less than 3 days from starting high dose GCs.
4. Diagnosis of active MAS confirmed by the treating rheumatologist, having ascertained the followings:

   a. Febrile subjects presenting with ferritin > 684 ng/mL. b. and any 2 of: i. Platelet count ≤ 181 x109/L ii. AST-level > 48 U/L iii. Triglycerides > 156 mg/dL iv. Fibrinogen level ≤ 360 mg/dL
5. Female subjects of child-bearing potential willing to use highly effective methods of contraception from study drug initiation to 6 months after the last dose of study drug.

   Specific inclusion criteria to Cohort 1 and Cohort 2
6. Cohort 1:

   1. Confirmed sJIA diagnosis. For subjects presenting with MAS in the context of the onset of sJIA, high presumption of sJIA will suffice for eligibility.
   2. Confirmed diagnosis of AOSD as per Yamaguchi criteria.
7. Cohort 2:

   1. Confirmed diagnosis of SLE as per SLICC'12 criteria.

Exclusion criteria

1. Primary HLH documented by either the presence of a known causative genetic mutation or abnormal perforin expression and CD107a degranulation assay as described with primary hemophagocytic lymphohistiocytosis or by the presence of family history.
2. Confirmed malignancy. Note: subjects with a suspected malignancy should have mononuclear cells typed by flow cytometry and/or tissue biopsy, as applicable, to rule out malignancy.
3. Treatment with canakinumab, JAK inhibitors, TNF inhibitors and tocilizumab at the time of emapalumab initiation.
4. Ongoing treatment with anakinra at a dose above 4 mg/kg at time of emapalumab initiation.
5. Subjects treated with etoposide for MAS in the last 1 month.
6. Clinically active mycobacteria (typical and atypical), Histoplasma Capsulatum, or Salmonella infections.
7. Evidence of leishmania infections.
8. Evidence of latent tuberculosis.
9. History of hypersensitivity or allergy to any component of the study drug.
10. Receipt of a Bacillus Calmette-Guerin (BCG) vaccine within 12 weeks prior to screening.
11. Receipt of a live or attenuated live (other than BCG) vaccine within 4 weeks prior to screening.
12. Pregnancy or lactating female subjects.

Ages: 6 Months to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2021-12-15 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2025-06-04 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects with complete response (CR) at Week 8 after first administration of emapalumab | 8 weeks
  Resolution of clinical signs and symptoms present at baseline: The MAS clinical activity will be measured on a visual analog scale (VAS) 10 cm.
  Resolution of clinical signs and symptoms present at baseline: The MAS clinical activity will be measured on a visual analog scale (VAS) 10 cm. Clinical signs will be considered as resolved if VAS is below or equal to 1/10.
  And
  Normalization of laboratory parameters relevant to MAS, as follows:
  WBC above LLN platelet count above LLN LDH below 1.5 ULN ALT below 1.5 ULN AST below 1.5 ULN fibrinogen higher than 100 mg/dL ferritin levels decreased by at least 80 % from values at screening or baseline (whichever is higher) or below 2000 ng/ml, whichever is low

SECONDARY OUTCOMES:
GCs tapering to a dose below 50% of prednisolone (PDN) equivalent at the time of emapalumab start or to the same (or lower) dose being administered before the occurrence of MAS whichever occurs first | At any time in the study, up to 1 year
  GC tapering as per investigator discretion
GCs tapering to ≤1mg/kg/day of PDN equivalent at any time during the study. | At any time in the study, up to 1 year
  GC tapering as per investigator discretion
Time to achieve GCs tapering as defined above. | At any time in the study, up to 1 year
  GC tapering as per investigator discretion
Time to first Complete Remission | At any time in the study, up to 1 year
  Time to CR
Proportion of subjects with overall response as defined by CR or PR | At any time in the study, up to 1 year
  Resolution of clinical signs and symptoms present at baseline: The MAS clinical activity will be measured on a visual analog scale (VAS) 10 cm.
Time to first overall response as defined by CR or PR | At any time in the study, up to 1 year
  CR defined as below:
  Resolution of clinical signs and symptoms present at baseline: The MAS clinical activity will be measured on a visual analog scale (VAS) 10 cm.
MAS recurrence at anytime after achievement of CR | At any time after CR, up to 1 year
  Time to MAS recurrence after CR
Withdrawal from the study due to lack of response as per Investigator decision | At any time in the study, up to 1 year
  Time to withdrawal
Survival time | At any time in the study, up to 1 year
  Time to Survival

OTHER OUTCOMES:
Adverse Events (AEs) (serious and non-serious). | At any time in the study, up to 1 year
  Incidence, severity, causality and outcomes of AEs
Study interruption due to safety reasons | At any time in the study, up to 1 year
  Number of subjects withdrawn due to safety reasons
Laboratory parameters | At any time in the study, up to 1 year
  Changes from baseline
Patient reported outcomes : PedsQL™; | Screening, Week 8, month 6 and 1 year
  Pediatric Quality of Life Inventory (PedsQL™; Generic Core Scales and Infant Scales, Acute versions)
Patient reported outcomes: Patient/Parent Global Impression of Severity | Screening, Week 8, month 6 and 1 year
  Health-related quality of life: Global Assessment: Patient/Parent Global Impression of Severity
Patient reported outcomes: Clinician Global Impression of Severity | Screening, Week 8, month 6 and 1 year
  Health-related quality of life: Global Assessment: Clinician Global Impression of Severity
PK endpoints | Every treatment visit until week 8, Day 60, Day 100, 6 months, 1 year
  Serum concentrations of emapalumab vs. time
PK endpoints CEOI, | Every treatment visit until week 8, Day 60, Day 100, 6 months, 1 year
  PK parameters by non-compartmental analysis: CEOI,
PK endpoints: λz, | Every treatment visit until week 8, Day 60, Day 100, 6 months, 1 year
  PK parameters by non-compartmental analysis: λz,
PK endpoints: CL, | Every treatment visit until week 8, Day 60, Day 100, 6 months, 1 year
  PK parameters by non-compartmental analysis: CL,
PK endpoints: Vss, | Every treatment visit until week 8, Day 60, Day 100, 6 months, 1 year
  PK parameters by non-compartmental analysis: Vss,
PK endpoints: MRTlast and MRTinf | Every treatment visit until week 8, Day 60, Day 100, 6 months, 1 year
  PK parameters by non-compartmental analysis: MRTlast and MRTinf, as applicable
PD endpoints per cohort: free IFN-γ and total IFNγ | Every treatment visit until week 8, Day 60, Day 100, 6 months, 1 year
  • Levels of circulating free IFN-γ at pre-dose, and total IFNγ (free IFN-γ+bound to emapalumab) after initiation of the study drug.
PD endpoints per cohort: chemokines | Every treatment visit until week 8, Day 60, Day 100, 6 months, 1 year
  Levels of the main IFN-γ-induced chemokines (CXCL9, CXCL10).
PD endpoints per cohort: sCD25) | Every treatment visit until week 8, Day 60, Day 100, 6 months, 1 year
  Levels of MAS markers (sCD25).
Immunogenicity endpoints | Treatment visit 1, week 8, 6 months, 1 year
  Occurrence of ADAs, Nab to emapalumab

CONTACTS AND LOCATIONS:
Overall Officials: Brian Jamieson, MD, Study Director — Swedish Orphan Biovitrum
Locations (44):
- United States (9):
  - UAB Hospital, Birmingham, Alabama
  - UCLA Health, Los Angeles, California
  - University of Florida, Gainesville, Florida
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - University of Minnesota Masonic Children's Hospital, Minneapolis, Minnesota
  - Akron Children's Hospital, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Nationwide Children's Hospital, Abigail Wexner Research Institute, Columbus, Ohio
  - UPMC Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
- Universitair Ziekenhuis Leuven, Leuven, Belgium
- Canada (5):
  - Alberta Children's Hospital, Calgary
  - University of Calgary, Calgary
  - Centre Hospitalier de l'Université de Montréal, Montreal
  - Centre Hospitalier Universitaire Sainte-Justine, Montreal
  - Hospital for sick children, Toronto
- China (3):
  - Beijing Children's Hospital, Beijing
  - Beijing Friendship Hospital, Beijing
  - Children's Hospital of Fudan University, Shanghai
- Czechia (2):
  - Fakultní nemocnice Olomouc, Olomouc
  - Vseobecna Fakultni Nemocnice v Praze, Prague
- France (4):
  - Hôpital Claude Huriez, Lille
  - Hôpital De La Conception, Marseille
  - Hôpital Necker-Enfants Malades, Paris
  - Hôpital Universitaire Pitié Salpêtrière, Paris
- Germany (2):
  - Charité Universitätsmedizin, Berlin
  - Universitätsklinikum Heidelberg, Heidelberg
- Italy (4):
  - IRCCS G. Gaslini, Genova
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan
  - Ospedale Pediatrico Bambino Gesù, Roma
  - IRCCS - Materno-Infantile Burlo Garofolo, Trieste
- Japan (4):
  - St. Marianna University School of Medicine Hospital, Kawasaki
  - Osaka Medical and Pharmaceutical University Hospital, Takatsuki
  - Tokyo Medical and Dental University Hospital, Tokyo
  - Yokohama City University Hospital, Yokohama
- UMC Utrecht, Utrecht, Netherlands
- Poland (3):
  - Szpital Specjalistyczny im. J. Dietla w Krakowie, Krakow
  - Wojewódzki Specjalistyczny Szpital Dziecięcy im. św. Ludwika w Krakowie, Krakow
  - Ortopedyczno - Rehabilitacyjny Szpital Kliniczny im. Wiktora Degi Uniwersytetu Medycznego im. Karola Marcinkowskiego w Poznaniu, Poznan
- Spain (4):
  - Hospital Sant Joan de Déu, Barcelona
  - Hospital Universitario La Paz, La Paz
  - Hospital Universitario, La Paz
  - Hospital Universitari i Politècnic La Fe, Valencia
- United Kingdom (2):
  - Great Ormond Street Hospital, London
  - Imperial College Healthcare NHS Trust, London

IPD SHARING:
Plan to Share IPD: No